CLINICAL TRIAL: NCT03448224
Title: The Development and Evaluation of a Behavioral Intervention to Reduce Indoor Tanning
Brief Title: Behavioral Intervention in Reducing Indoor Tanning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jerod L Stapleton, PhD (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Jerod L Stapleton, PhD, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 131315; NCI-2018-00063 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Pro2013003349 (Other: Rutgers Cancer Institute of New Jersey); 131315 (Other: Rutgers Cancer Institute of New Jersey); K07CA175115 (NIH); P30CA072720 (NIH)
Record Dates: First submitted 2018-02-02; First posted 2018-02-28 (Actual); Results first posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-09

CONDITIONS: Healthy Subject

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (web-based Indoor Tanning intervention) (Experimental): Participants receive intervention, weekly text messages about IT reduction, and personalized booster intervention. Participants then receive text messages twice weekly for 4 weeks.
  Interventions: Other: Questionnaire Administration; Other: Internet-Based Intervention
- Group II (wait-list) (Active Comparator): Participants are placed on wait-list and may receive full intervention after follow-up.
  Interventions: Other: Questionnaire Administration

INTERVENTIONS:
Other: Questionnaire Administration — Questionnaire
Other: Internet-Based Intervention — Intervention
  Arms: Group I (web-based Indoor Tanning intervention)

SUMMARY:
This randomized clinical trial tests the efficacy of a behavioral intervention works in reducing indoor tanning. Artificial ultraviolet indoor tanning increases the chance of developing skin cancers. Behavioral interventions use techniques to help participants change the way they react to environmental triggers that may cause a negative reaction.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

To develop and evaluate an online tailored indoor tanning (IT) intervention based on findings from phase 1.

OUTLINE:

INTERVENTION: Participants are randomized to 1 of 2 groups.

GROUP I: Participants receive intervention, weekly text messages about IT reduction, and personalized booster intervention. Participants then receive text messages twice weekly for 4 weeks.

GROUP II: Participants are placed on wait-list and may receive full intervention after follow-up.

After completion of study, patients are followed up at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Use of IT at least 25 times in the past year
* Women

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 54 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2019-02-06 (Actual); Study Completion 2019-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerod Stapleton, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stapleton JL, Ray AE, Glenn SD, McLouth LE, Parmar V, Manne SL. A randomized controlled trial of a web-based personalized feedback intervention targeting frequent indoor tanning bed users: Engagement, acceptability, and preliminary behavioral outcomes. J Health Psychol. 2022 Mar;27(4):923-935. doi: 10.1177/1359105320982038. Epub 2020 Dec 22. PMID 33353412

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Qualtrics Sample Providers emailed advertisements for an online screening survey to members of internet panels and posted online advertisements. Recruitment flyers with contact information were posted on campus and in classrooms and on internet ads on social media and Craigslist. Baseline assessments were completed between April and November 2018
Pre-assignment Details: One participant removed after assignment because of failed quality check with baseline data.
Groups:
- Group II (Wait-list): Participants are placed on wait-list and receive full intervention after follow-up.
  Questionnaire Administration: Questionnaire
Period: Overall Study
Arm/Group | Group I (Web-based Indoor Tanning Intervention) | Group II (Wait-list)
Started | 28 | 26
Completed | 27 | 26
Not Completed | 1 | 0
Not completed — Provided same answer to every question | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I (Web-based Indoor Tanning Intervention) | Group II (Wait-list) | Total
Number analyzed (Participants) | 27 | 26 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 26 | 53
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.88 (1.66) | 22.29 (2.05) | 22.60 (1.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 26 | 53
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 22 | 23 | 45
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Customized: Causasian/White | 24 | 21 | 45
  Race: Customized: Black or African American | 1 | 2 | 3
  Race: Customized: Other | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Prior 2-Month Indoor Tanning Sessions Reported by Participants on a Follow-up Survey
Description: On the follow-up assessment administered 3 months after the baseline assessment, participants will estimate the number of times they used a tanning bed or booth with tanning lamps in the past 2 months with an open-ended response.
Time Frame: Up to 3 months
Measure: Mean (Standard Deviation); unit: indoor tanning sessions
Arm/Group | Group I (Web-based Indoor Tanning Intervention) | Group II (Wait-list)
Number analyzed (Participants) | 27 | 26
indoor tanning sessions | 11.5 (2.1) | 7.9 (2.1)

2. Secondary Outcome: Perceived Difficulty (Self-efficacy) in Quitting Tanning
Description: Measured at post-intervention data collection (3 months post intervention) using single item assessment: "How hard would it be for you to stop using tanning beds/booths?" (Please answer on a scale for 0-10, where 0 is "Not at all hard", 10 is "Extremely hard").
Time Frame: At 3 months post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group I (Web-based Indoor Tanning Intervention) | Group II (Wait-list)
Number analyzed (Participants) | 27 | 26
score on a scale | 5.0 (0.6) | 5.0 (0.6)

3. Secondary Outcome: Sunburns
Description: On the follow-up assessment administered 3 months after the baseline assessment, participants will estimate the number of times they had a sunburn in the past 2 months with an open-ended response.
Time Frame: Up to 3 months
Measure: Mean (Standard Deviation); unit: sunburns
Arm/Group | Group I (Web-based Indoor Tanning Intervention) | Group II (Wait-list)
Number analyzed (Participants) | 27 | 26
sunburns | 1.9 (0.4) | 1.1 (0.4)

4. Secondary Outcome: Intentions to Use Indoor Tanning
Description: For tanning intentions, participants indicated how likely they were to use an indoor tanning bed in the next year on a 6-point response scale anchored with 1 = Extremely unlikely and 6 = Extremely likely
Time Frame: Up to 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group I (Web-based Indoor Tanning Intervention) | Group II (Wait-list)
Number analyzed (Participants) | 27 | 26
score on a scale | 5.0 (0.3) | 4.8 (0.3)

5. Secondary Outcome: Number of Participants Expressing Positive Interest in Changing Tanning
Description: Interest in changing tanning was assessed using a single item: Would you like to reduce or quit indoor tanning if you could do so easily? Responses coded as 0 = no and 1 = yes
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Web-based Indoor Tanning Intervention) | Group II (Wait-list)
Number analyzed (Participants) | 27 | 26
Participants | 18 | 12

ADVERSE EVENTS:
Time Frame: The time frame from over which potential adverse events data were collected was during the intervention (duration of four weeks) through the time until follow-up data was collected (3 months post intervention) for a total of 4 months of observation for adverse events for each participant.
Description: The definition does not differ.
Arm/Group | Group I (Web-based Indoor Tanning Intervention) | Group II (Wait-list)
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/26
Other Adverse Events (participants affected / at risk) | 0/27 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2019-01-25): https://cdn.clinicaltrials.gov/large-docs/24/NCT03448224/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-01-25): https://cdn.clinicaltrials.gov/large-docs/24/NCT03448224/Prot_SAP_001.pdf